CLINICAL TRIAL: NCT03741634
Title: Shamba Maisha: Assessing the Preliminary Effects of a Multisectoral Agricultural Intervention on the Sexual and Reproductive Health of HIV-affected Adolescent Girls in Western Kenya
Brief Title: Assessing the Preliminary Effects of a Multisectoral Agricultural Intervention on Adolescent Girls' Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Kenya Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R21HD095739 (NIH)
Record Dates: First submitted 2018-11-07; First posted 2018-11-15 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Adolescent Behavior; Sexual Behavior; Reproductive Behavior
Keywords: adolescent health; sexual health; reproductive health; food security
MeSH Terms: conditions — Adolescent Behavior; Sexual Behavior; Reproductive Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants enrolled at one study location will receive the Multi-sectoral agricultural intervention as specified below under the intervention.
  Interventions: Other: Multi-sectoral agricultural intervention
- No intervention (No Intervention): During the study, participants enrolled at one study location will non receive the Multi-sectoral agricultural intervention. At the end of the study, participants in this arm will be eligible for education in financial management and sustainable farming practices and those who pay the loan down payment will be eligible for a small loan to purchase a human-powered water pump, seeds, fertilizers and, pesticides.

INTERVENTIONS:
Other: Multi-sectoral agricultural intervention — Adult participants in the intervention arm receive a loan (~$175) from a well-established Kenyan bank used to get a human-powered water pump, seeds, fertilizers and, pesticides, and education in financial management and sustainable farming practices.
  Arms: Intervention

SUMMARY:
The goal of this study is to understand how the Shamba Maisha household agricultural and economic intervention impacts the sexual, reproductive, and nutritional health of adolescent girls. The intervention includes: a) a human-powered water pump and other required farm commodities, b) a micro-finance loan (~$75) to purchase the pump and agricultural implements, and c) education in sustainable farming practices.

DETAILED DESCRIPTION:
Food insecurity (FI) and poverty are important drivers of HIV vulnerability among adolescent girls, and contribute to worse sexual and reproductive health (SRH) outcomes. While most approaches to improving adolescent SRH outcomes have focused on individual-centered approaches alone, integrated family-level interventions that address the underlying context for risk behaviors such as poverty and FI may be more effective in reducing adverse SRH outcomes. A household-level multisectoral agricultural and finance intervention in Nyanza Region, Kenya called Shamba Maisha (SM) designed to mitigate household FI and improve health in HIV-affected households has been successfully developed and piloted. In mid-2016, a large cluster-randomized controlled trial (RCT) of SM was launched, targeting 704 adults and 352 young children to test the effectiveness of this intervention. This pilot study leverages the SM RCT infrastructure to recruit up to 240 adolescent girls residing in SM households and assess the impact of the SM intervention at the household level on adolescent girls' SRH outcomes at study endline. The central hypothesis is that improvements in household FI and wealth will contribute to reduced sexually transmitted infections (STIs), HIV, and unintended pregnancies among adolescent girls. To test this hypothesis, demographic, behavioral, clinical, and biological data from adolescent girls and their caregivers living in intervention and control SM households will be collected. The primary outcomes are food security, depressive symptoms, and sexual risk behaviors in the adolescent girls. The secondary outcomes are pregnancy/unintended pregnancy, HIV, herpes simplex virus 2 (HSV-2), and nutritional status in the adolescent girl.

The ultimate goal is to develop an intervention tailored specifically to the needs of adolescent girls to help reverse the cycle of FI, poverty, low empowerment, and poor SRH outcomes among adolescent girls. If proven efficacious, the proposed intervention may: 1) halt or slow down the cycle of incident HIV, other STIs, and unintended pregnancies to improve the lives of adolescent girls in similar settings, and 2) help achieve several top Sustainable Development Goals (SDG) including SDG 1 (zero poverty), SDG 2 (zero hunger), SDG 3 (good health and wellbeing), and SDG 5 (gender equality).

ELIGIBILITY:
Inclusion Criteria:

* an adult participating in the parent study
* a currently unmarried adolescent girl aged 13-20 years old (preferred target of 15-19)
* the adolescent girl has a parent/primary guardian age >18 years old who resides in the household

Exclusion Criteria:

* adolescent girls with a confirmed HIV diagnosis by clinical records prior to the start of SM
* married adolescent girls
* those who do not speak Dholuo, Swahili, or English
* those who are heads of households
* those ages 18 to 20 who are enrolled in the parent study
* those with inadequate cognitive and/or hearing capacity.

Ages: 13 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 241 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Food insecurity | Endline / 2 years
  Food insecurity as assessed by the Household Food Insecurity Access Scale (HFIAS; score range 0-27 [least to most food insecure]).
Depressive symptoms | Endline / 2 years
  Depression, assessed by the 15 item Hopkins Symptom Checklist-Depression (score range 1-4 [least to most depressed].
Unprotected sex | Endline / 2 years
  Percentage of time not used condoms over past six months

SECONDARY OUTCOMES:
Percentage of participants who become pregnant | Endline / 2 years
  Measured by urine pregnancy test
Unintended pregnancy | Endline / 2 years
  Unintended pregnancy as assessed by the London Measure of Unplanned Pregnancy
HIV | Endline / 2 years
  Serial rapid HIV tests based on the Kenyan Ministry of Health guidelines
HSV-2 | Endline / 2 years
  HSV-2 by Kalon assay (Herpes Simplex Type 2 IgG ELISA, Kalon Biologics, Ltd.)
Body mass index-for-age-Z-score | Endline / 2 years
  Weight and height will be combined to report BMI in kg/m^2 as Z score
Physical health | Endline / 2 years
  Assessed by the Medical Outcomes Study Short Form (SF-36, score range 0-100 [poor to excellent health])
Number of sexual partners | Endline / 2 years
  Number of sexual partners over past six months

OTHER OUTCOMES:
Anxiety | Endline / 2 years
  Measured by the Generalized Anxiety Disorder Scale (GAD-7, 0-21 [least to most anxious]).
Empowerment | Endline / 2 years
  Measured by the Child and Youth Resilience Measure (CYRM-12, score range 12-60 [least to most resilient]).
School attendance | Endline / 2 years
  Days of school missed in previous term

CONTACTS AND LOCATIONS:
Overall Officials: Sheri D Weiser, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (16):
- Kenya (16):
  - Kitare, Suba, Homa Bay County
  - Sindo, Suba, Homa Bay County
  - Muhuru Bay, Nyatike, Migori County
  - Sori Lakeside, Nyatike, Migori County
  - Minyenya, Rongo, Migori County
  - Ngode, Rongo, Migori County
  - Oyani, Rongo, Migori County
  - Nyamasare, Uriri, Migori County
  - Hongo Ogosa, Kisumu
  - Kisumu District Hospital, Kisumu
  - Lumumba, Kisumu
  - Nyangande, Kisumu
  - Osingo, Kisumu
  - Pandiperi, Kisumu
  - Railways, Kisumu
  - Suna Ragana, Migori

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pandit JA, Sirotin N, Tittle R, Onjolo E, Bukusi EA, Cohen CR. Shamba Maisha: a pilot study assessing impacts of a micro-irrigation intervention on the health and economic wellbeing of HIV patients. BMC Public Health. 2010 May 11;10:245. doi: 10.1186/1471-2458-10-245. PMID 20459841
- [Background] Zakaras JM, Weiser SD, Hatcher AM, Weke E, Burger RL, Cohen CR, Bukusi EA, Dworkin SL. A Qualitative Investigation of the Impact of a Livelihood Intervention on Gendered Power and Sexual Risk Behaviors Among HIV-Positive Adults in Rural Kenya. Arch Sex Behav. 2017 May;46(4):1121-1133. doi: 10.1007/s10508-016-0828-x. Epub 2016 Aug 9. PMID 27507020
- [Background] Weiser SD, Bukusi EA, Steinfeld RL, Frongillo EA, Weke E, Dworkin SL, Pusateri K, Shiboski S, Scow K, Butler LM, Cohen CR. Shamba Maisha: randomized controlled trial of an agricultural and finance intervention to improve HIV health outcomes. AIDS. 2015 Sep 10;29(14):1889-94. doi: 10.1097/QAD.0000000000000781. PMID 26214684
- [Background] Cohen CR, Steinfeld RL, Weke E, Bukusi EA, Hatcher AM, Shiboski S, Rheingans R, Scow KM, Butler LM, Otieno P, Dworkin SL, Weiser SD. Shamba Maisha: Pilot agricultural intervention for food security and HIV health outcomes in Kenya: design, methods, baseline results and process evaluation of a cluster-randomized controlled trial. Springerplus. 2015 Mar 12;4:122. doi: 10.1186/s40064-015-0886-x. eCollection 2015. PMID 25992307
- [Derived] Onono MA, Frongillo EA, Sheira LA, Odhiambo G, Wekesa P, Conroy AA, Cohen CR, Bukusi EA, Weiser SD. Links between Household-Level Income-Generating Agricultural Intervention and the Psychological Well-Being of Adolescent Girls in Human Immunodeficiency Virus-Affected Households in Southwestern Kenya: A Qualitative Inquiry. J Nutr. 2023 Dec;153(12):3595-3603. doi: 10.1016/j.tjnut.2023.10.008. Epub 2023 Oct 18. PMID 37863268
- See also: Shamba Maisha study website — https://shambamaisha.ucsf.edu/